CLINICAL TRIAL: NCT03634098
Title: Identification and Validation of Noninvasive Biomarkers (Virtual Biopsy) of the Diagnosis and Severity of NASH in Type 2 Diabetics: a Cross-sectional Study
Brief Title: Identification and Validation of Noninvasive Biomarkers of the Diagnosis and Severity of NASH in Type 2 Diabetics
Acronym: Quid-Nash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: P171105j; 2018-A00311-54 (Other: IDRCB)
Record Dates: First submitted 2018-07-16; First posted 2018-08-16 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-03

CONDITIONS: Type2 Diabetes
Keywords: Patients
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Volunteers (Experimental): Exams performed on volunteers with other purpose than liver disease or diabetes in two centers:
  * MRI
  * Ultrasound AixPlorer These examinations are carried out in 2 differents centers at 1month intervals
  Interventions: Device: new quantitative imaging techniques with contast products
- T2D liver test abnormalities's participants (Experimental): Exams performed on type 2 diabetic patients with liver test abnormalities :
  * sample for analysis and biocollection
  * MRI +/-Primovist
  * Ultrasound AixPlorer +Sonovue
  Interventions: Device: new quantitative imaging techniques with contast products; Diagnostic Test: blood sample; Diagnostic Test: second generation tests
- T2D participants without liver test abnormality (No Intervention): type 2 diabetic participants without liver test abnormality and not undergoing liver biopsy

INTERVENTIONS:
Device: new quantitative imaging techniques with contast products — magnetic resonance +/- Primovist and ultrafast ultrasound UFUS +Sonovue
  Arms: T2D liver test abnormalities's participants; Volunteers
Diagnostic Test: blood sample — extensive clinical-biological phenotyping data; and / or data obtained by different omic approaches (metabolomics, targeted genetics, transcriptomics). Extracellular vesicle and immune cell profiling will complement this data
  Arms: T2D liver test abnormalities's participants
Diagnostic Test: second generation tests — second generation tests NIT-NASHr et NIT-A2F2
  Arms: T2D liver test abnormalities's participants

SUMMARY:
Metabolic diseases of the liver are silent affections whose morbidity is important. About 70% of patients with type 2 diabetes (T2D) are concerned. Of these, 50% develop clinically significant lesions (including non-alcoholic steatohepatitis or NASH) as they are associated with an increased risk of complications; and 15% progress to severe fibrosis or cirrhosis. These diseases are slowly progressive and asymptomatic. Their pathophysiology is poorly known. Management is hampered by the absence of a specific diagnostic marker, the need for invasive diagnostic procedures (liver biopsy), and the lack of established treatment.

QUID-NASH aims to develop a virtual liver biopsy in T2D participants, based on the identification of single or combined, multimodal, non-invasive biomarkers obtained by new quantitative imaging techniques (magnetic resonance and ultrafast ultrasound UFUS); and /or extensive clinical-biological phenotyping data; and/or data obtained by different omic approaches (metabolomics, targeted genetics, transcriptomics). Extracellular vesicle and immune cell profiling will complement these phenotyping data. This approach will also enable us to improve our understanding of pathophysiology (new signaling pathways, new therapeutic targets).

DETAILED DESCRIPTION:
Metabolic diseases of the liver are silent affections whose morbidity is important. About 70% of patients with type 2 diabetes (T2D) are concerned. Of these, 50% develop clinically significant lesions (including non-alcoholic steatohepatitis or NASH) as they are associated with an increased risk of complications; and 15% progress to severe fibrosis or cirrhosis. These diseases are slowly progressive and asymptomatic. Their pathophysiology is poorly known. Management is hampered by the absence of a specific diagnostic marker, the need for invasive diagnostic procedures (liver biopsy), and the lack of established treatment. Non-invasive methods ("first-generation" tests) have recently seen significant growth: commercialization of FibroTest as a marker of fibrosis; FibroTest, Fibrometer and FibroScan, for the initial assessment of adult chronic hepatitis C; FibroTest, Fibrometer, and Enhanced Liver Fibrosis test (ELF-test) for diagnosis of metabolic liver disease and diagnosis of fibrosis; SteatoTest (APHP patent) for the diagnosis of steatosis. The ActiTest (APHP patent) is widely used in evaluating the necrotic-inflammatory activity of chronic viral hepatitis C and B. For the diagnosis of NASH alone the ActiTest is validated. The NashTest (APHP patent) is little used. Several biomarkers of imaging (liver ultrasound, FibroScan Controller Attenuated Parameter (CAP), elastography and nuclear magnetic resonance) are widely used for the diagnosis of steatosis. Two new "second generation" blood tests (APHP patents) are under development, Non Invasive Test-NASHr (NIT-NASHr), and NIT-A2F2. NIT-NASHr is a new combination of the components of SteatoTest and NASH-Test to assess the severity of NASH. NIT-A2F2 is a combination of NIT-NASHr and FibroTest for the diagnosis of clinically significant liver metabolic disease. These tests will be the subject in the project of a validation of their performances in the context of use (T2D without other liver disease). At the same time, significant progress has been made in integrating omic data to characterize various pathologies and to identify their mechanisms. The transcriptomics and metabolomics of body fluids are particularly promising for the construction of "third generation" tests.

QUID-NASH aims to develop a virtual liver biopsy in T2D participants, based on the identification of single or combined, multimodal, non-invasive biomarkers obtained by new quantitative imaging techniques (magnetic resonance and ultrafast ultrasound UFUS); and / or extensive clinical-biological phenotyping data; and / or data obtained by different omic approaches (metabolomics, targeted genetics, transcriptomics). Extracellular vesicle and immune cell profiling will complement this data. This approach will also enable us to improve knowledge of the pathology (new signaling pathways, new therapeutic targets).

ELIGIBILITY:
Pilot phase : Volunteers (for reproducibility study) Inclusion criteria

* Voluntary
* Person aged 18 or over

Criteria for non-inclusion

* Refusal or inability to sign consent
* Vulnerable person according to article L1121-6 of the CSP
* Protected person of age

Clinical Study of Clinically Significant NASH or NASH Markers Performance with Standard NASH Criteria (patient with liver biopsy) Inclusion criteria

* Participant aged 18 or over
* Diabetic type 2 (ADA / WHO criteria mentioned in section 20.5)
* Liver biopsy planned in day hospital (HDJ) as part of routine care (indication of biopsy: or ALT> 30 IU for men or> 20 IU for women less than 1 month old) and/or steatosis on ultrasound )
* Hemoglobin> 7g / dL (or> 10 g / dL in case of cardiovascular or respiratory pathology)

Criteria for non-inclusion

* Refusal or inability to sign consent
* Vulnerable person: person deprived of liberty by a judicial or administrative decision, or subject to psychiatric care, and person admitted to a health or social institution for purposes other than that of research
* Protected person of age
* No affiliation or non-beneficiary of a social security scheme
* Pregnant or lactating woman
* Contraindication to MRI according to the French Society of Radiology (mentioned in section 20.4)
* Corpulence incompatible with the realization of an MRI
* Disease related to other etiologies

  * Alcoholic liver disease
  * Current infection of hepatitis B virus
  * Current infection of hepatitis C virus
  * Autoimmune hepatitis according to AASLD and EASL oTransferrin saturation>50%
  * Alpha-1 antitrypsin deficiency ZZ or SZ
  * Wilson's disease
  * Obstruction of the blood vessels or bile ducts on ultrasound (on routine ultrasound If nothing is mentioned on the report, it is considered that there is no obstruction of the vessels blood or bile ducts)
* Liver transplant

Subgroup with Primovist:

-Contraindication to gadoxetic acid: Hypersensitivity to gadoxetic acid or to one of the excipients depending on the composition. Severe renal faillure (GFR <30 mL / min / 1.73 m²).

Subgroup with Sonovue:

-Any contraindication to Sonovue®, namely: hypersensitivity to sulfur hexafluoride or to one of the excipients of the specialty, right-left shunt, severe pulmonary arterial hypertension (> 90 mmHg), uncontrolled systemic hypertension, respiratory distress syndrome in adults, combination with dobutamine

Clinical study of the performance of second-generation tests for the diagnosis of metabolic liver disease: border population Inclusion criteria

* Consecutive patients aged 18 years or over
* Diabetic Type 2 (ADA / WHO criteria mentioned in section 20.5)

Criteria for non-inclusion

* Refusal or inability to sign consent
* Vulnerable person: person deprived of liberty by a judicial or administrative decision, person under psychiatric care and person admitted to a health or social institution for purposes other than research
* Protected person of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 970 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
To study in type 2 diabetic participants with liver biopsy, the performance of a composite biomarker (3rd generation test) for the diagnosis of NASH | 1 month
  Histological diagnosis of NASH (as established by centralized re-reading of liver biopsy slides), blinded to omic results and imaging.

SECONDARY OUTCOMES:
To study in type 2 diabetic participants with or without liver biopsy, performance of a composite biomarker for the diagnosis of clinically significant metabolic liver diseases | 1 month
  diagnosis of clinically significant liver metabolic disease (SAF-Score ≥A2 or ≥F2) adjudicated by an independent committee
To study in type 2 diabetic participants with liver biopsy, the performance of a single or composite biomarker for the diagnosis of NASH elemental lesions | 1 month
  histological diagnosis of elementary lesions of NASH (lobular inflammation, ballooning, steatosis)
To study inter-center and intra-participants reproducibility of imaging measurements. a graphical evaluation will be conducted using a representation of Bland-Altman. | 1 month
  By MRI: steatosis, biomechanical properties, T1, diffusivity
To study inter-center and intra-participants reproducibility of imaging measurements.a graphical evaluation will be conducted using a representation of Bland-Altman. | 1 month
  By AixPlorer ultrasound: steatosis, biomechanical properties, vascular properties
To study in type 2 diabetic participants the performance of second-generation tests for the diagnosis of metabolic liver diseases | 1 day
  metabolic liver disease (adjudicated by an independent committee)
Constitution of a bio-collection | 1 month
  stool
Constitution of a bio-collection | 1 month
  urine
Constitution of a bio-collection | 1 month
  plasma
Constitution of a bio-collection | 1 month
  serum
Constitution of a bio-collection | 1 month
  mononuclear cells of peripheral blood
Constitution of a bio-collection | 1 month
  Liver tissue

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Castera, Principal Investigator — APHP
Locations (1):
- Hôpital Beaujon, Clichy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Castera L, Garteiser P, Laouenan C, Vidal-Trecan T, Vallet-Pichard A, Manchon P, Paradis V, Czernichow S, Roulot D, Larger E, Pol S, Bedossa P, Correas JM, Valla D, Gautier JF, Van Beers BE; QUID NASH investigators. Prospective head-to-head comparison of non-invasive scores for diagnosis of fibrotic MASH in patients with type 2 diabetes. J Hepatol. 2024 Aug;81(2):195-206. doi: 10.1016/j.jhep.2024.03.023. Epub 2024 Mar 27. PMID 38548067
- [Derived] Poynard T, Deckmyn O, Peta V, Paradis V, Gautier JF, Brzustowski A, Bedossa P, Castera L, Pol S, Valla D; Quid-Nash Consortium. Prospective direct comparison of non-invasive liver tests in outpatients with type 2 diabetes using intention-to-diagnose analysis. Aliment Pharmacol Ther. 2023 Nov;58(9):888-902. doi: 10.1111/apt.17688. Epub 2023 Aug 29. PMID 37642160
- [Derived] Poynard T, Paradis V, Mullaert J, Deckmyn O, Gault N, Marcault E, Manchon P, Si Mohammed N, Parfait B, Ibberson M, Gautier JF, Boitard C, Czernichow S, Larger E, Drane F, Castille JM, Peta V, Brzustowski A, Terris B, Vallet-Pichard A, Roulot D, Laouenan C, Bedossa P, Castera L, Pol S, Valla D; Quid-Nash consortium. Prospective external validation of a new non-invasive test for the diagnosis of non-alcoholic steatohepatitis in patients with type 2 diabetes. Aliment Pharmacol Ther. 2021 Oct;54(7):952-966. doi: 10.1111/apt.16543. Epub 2021 Aug 16. PMID 34398492